CLINICAL TRIAL: NCT05597527
Title: A Single Arm, Exploratory, Multicenter Clinical Study of Fluzopari Combined With Apatinib Neoadjuvant Therapy in Patients With Advanced Non R0 Resectable Ovarian Cancer
Brief Title: Fluzopari Combined With Apatinib for the Neoadjuvant Treatment of Unresectable Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPing
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Cancer
Keywords: Fluzopari; Apatinini
MeSH Terms: conditions — Ovarian Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzopari and Apatinib group (Experimental): Fluzopari and Apatinib were used in patients with newly diagnosed ovarian cancer before any treatment. The daily dose should be strictly controlled according to the experimental design.
  Interventions: Drug: Fluzopari and apatinib

INTERVENTIONS:
Drug: Fluzopari and apatinib — Fluzopari was used as 100mg capsules orally twice a day (one time in the morning and one time in the evening), every four weeks as a cycle, a total of 3-4 cycles. Apatinib was used as 250 mg orally once a day, every 4 weeks as a cycle, 2-3 cycles in total, and stop 4 weeks before operation.

SUMMARY:
This is a single arm, multi center, exploratory clinical study to evaluate the efficacy and safety of fluzoparide combined with alpatinib as neoadjuvant therapy in patients with BRCA1/2 gene mutation or HRD gene mutation, advanced ovarian cancer, primary peritoneal cancer, fallopian tube cancer ((FIGO stage III or IV), who can not achieve R0 tumor reduction surgery after imaging evaluation or laparoscopic evaluation .

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged between 18 and 75 years old;
2. Patients received open surgery, laparoscopic surgery, or coarse needle aspiration biopsy and confirmed as high-grade serous or endometrioid ovarian cancer, peritoneal cancer, or fallopian tube cancer (hereinafter referred to as ovarian cancer). FIGO stage III-IV;
3. BRCA1/2 gene mutation or HRD gene mutation is confirmed by testing tissue or blood samples;
4. According to RECIST 1.1 standard, the patient has at least one target lesion with measurable diameter (the long diameter of CT scan for tumor lesions is ≥ 10mm, the short diameter of CT scan for lymph node lesions is ≥ 15mm, and the scanning thickness is 5mm);
5. Judge the patients who cannot achieve R0 tumor reduction or cannot tolerate surgery. The criteria for failing to achieve R0 tumor reduction include but are not limited to:

(1) Fagotti score ≥ 8; (2) When the laparoscopic evaluation method is difficult to implement, the upper abdomen CT score is ≥ 3 (SUDANCT score);

The criteria for surgical intolerance are as follows:

(3) Body mass index: BMI ≥ 40.0; (4) Various chronic diseases; (5) Malnutrition or hypoproteinemia; (6) Moderate to massive ascites; 6. ECOG PS 0-1 point; 7. The main organs function normally and meet the following standards:

1. The blood routine examination standard shall meet: (no blood transfusion within 14 days)

   1. HB≥100g/L，
   2. WBC≥3 × 109/L
   3. ANC≥1.5 × 109/L，
   4. PLT≥100 × 109/L；
2. Biochemical examination shall meet the following standards:

   1. BIL ≤ 1.5 times the upper limit of normal value (ULN);
   2. ALT and AST ≤ 2.5 × ULN, ALT and AST ≤ 5 in patients with liver metastasis × ULN；
   3. Serum Cr ≤ 1.5 × ULN。 8. International normalized ratio (INR) OR prothrombin time (PT), activated partial thrombin activity time (aPTT) ≤ 1.5 × ULN, unless the patient is receiving anticoagulant treatment, as long as PT or aPTT is within the expected treatment range of anticoagulant drugs; 9. There is no obstacle of strict center of gravity, lung, liver and kidney; 10. Women of childbearing age must have a pregnancy test (serum) within 7 days before enrollment, and the result is negative, and are willing to use appropriate methods of contraception during the test period and 8 weeks after the last administration of the test drug; 11. Estimated total survival time ≥ 6 months, postoperative survival time ≥ 3 months; 12. Sign the written informed consent, and be able to comply with the visit and relevant procedures specified in the scheme.

Exclusion Criteria:

1. Other clinical drug experiments in which other experimental research drugs are used together with the study;
2. In addition to this study, use other cancer neoadjuvant therapies, including but not limited to chemotherapy, radiotherapy, targeted therapy, immunotherapy, microbial therapy, traditional Chinese medicine therapy and other experimental treatments;
3. Patients known to be allergic to fluzoparide or allergic to active or non active components of fluzoparide with similar chemical structure;
4. Patients known to be allergic to appatinib or allergic to active or inactive components of drugs with similar chemical structure to appatinib;
5. It is impossible to swallow the oral drug and any gastrointestinal disease that may interfere with the absorption and metabolism of the study drug, such as uncontrollable nausea and vomiting, gastrointestinal obstruction or malabsorption;
6. Have used known or possible PARP inhibitors and anti vascular production inhibitors in the past;
7. Symptomatic or uncontrolled brain metastasis requiring simultaneous treatment, including but not limited to surgery, radiotherapy and/or corticosteroids, or clinical manifestations of spinal cord compression;
8. Subjects suffered from other malignant diseases in the past 3 years, except skin squamous cell carcinoma, basal like carcinoma, breast intraductal carcinoma in situ or cervical carcinoma in situ;
9. The patient was previously or currently diagnosed as myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
10. Recently (within 3 months), there has been intestinal obstruction and gastrointestinal perforation;
11. There are clinical cardiac symptoms or diseases that are not well controlled, such as: (1) NYHA level 2 or above cardiac insufficiency (2) unstable angina pectoris (3) acute myocardial infarction within one year (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention (5) QTc>470ms;
12. Any bleeding event with a severe grade of 2 or above in CTCAE 5.0 occurred within 4 weeks before the first trial medication;
13. People with hypertension who can not be well controlled after antihypertensive drug treatment (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
14. Idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, organized pneumonia, drug pneumonia, or active pneumonia shown on CT during screening period have been or are currently present;
15. Those with abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4s), who have bleeding tendency or are receiving thrombolytic or anticoagulant treatment (including but not limited to patients requiring long-term anticoagulant treatment), are allowed to receive low dose low molecular weight heparin or oral aspirin preventive anticoagulant treatment during the trial;
16. Diagnose patients with deep vein thrombosis (except intermuscular vein thrombosis);
17. People with a history of hereditary or acquired haemorrhagic disease or blood coagulation dysfunction. There were bleeding symptoms with significant clinical significance or clear bleeding tendency within 3 months before the first trial drug use, such as gastrointestinal bleeding, bleeding gastric ulcer, etc;
18. The subject has congenital or acquired immune deficiency (such as HIV infected persons), or active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA ≥ 500 IU/ml; hepatitis C reference: HCV antibody positive and HCV copy number>the upper limit of normal value);
19. The patient received platelet or red blood cell infusion within four weeks before the start of the study drug treatment;
20. Patients who are pregnant or nursing, or who plan to become pregnant during the study treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 3-month
  The percentage of patients received R0 resection after Fluzopari and Apatinib neoadjuvant treatment.
Overall Response Rate (ORR) | 3-month
  ORR is defined as the proportion of participants achieving Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST (v.1.1). Per RECIST 1.1, CR is defined as the disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of diameters (SoD) of target lesions.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 3-month
  Disease control rate is defined as the proportion of participants achieving Complete Response (CR), Partial Response (PR) or Stable Disease (SD) according to RECIST1.1.
Complete pathologic response rate(CPR) | 3-month
  Complete pathologic response rate is measured according to Miller-Panye system.
Progression Free Survival (PFS) | 3-year
  PFS is defined as the time in months from the date of first study drug administration to the date of first documentation of progressive disease (PD) or death as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Overall survival (OS) | 5 years
  OS is defined as the time from the study enrollment to death due to any cause.
Incidence rate of adverse events | 5 years
  The ratio of the number of cases with adverse events to the total number of cases available for evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Lin An, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No